CLINICAL TRIAL: NCT02179138
Title: EVALUATION OF A USER-FILLED, PAPER APPLICATOR FOR DELIVERY OF TENOFOVIR 1% GEL AMONG WOMEN IN RURAL KWAZULU-NATAL, SOUTH AFRICA
Brief Title: Paper Applicator Acceptability Study
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study no longer relevant based on change in regulatory pathway for TFV 1% gel
Sponsor: CONRAD (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CAPRISA 070
Record Dates: First submitted 2014-06-27; First posted 2014-07-01 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: HIV Prevention
MeSH Terms: interventions — Gels

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TFV 1% Gel (Other): TFV 1% gel with the user-filled paper applicator
  Interventions: Drug: TFV 1% gel

INTERVENTIONS:
Drug: TFV 1% gel

SUMMARY:
To assess the acceptability of a user-filled, paper, applicator for delivery of tenofovir (TFV) gel among women at high risk of acquiring human immunodeficiency virus (HIV) in rural KwaZulu-Natal, South Africa.

DETAILED DESCRIPTION:
CAPRISA 070 is designed to enroll rural women who exit from CAPRISA 008 - an ongoing trial assessing implementation, effectiveness and safety of TFV gel in KwaZulu-Natal, South Africa. All study participants in CAPRISA 008 have also participated in CAPRISA 004 and thus have several years of experience using TFV gel with the prefilled, plastic applicator. CAPRISA 070 will allow us to assess acceptability of the user-filled, paper applicator among women who have had extensive experience with the pre-filled, plastic applicator and are well-positioned to provide feedback and comparisons on a new gel delivery method.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Women who previously participated in CAPRISA 008
* Able and willing to provide first person informed consent to be screened for, and to enroll in, the study
* Allow access to their CAPRISA 008 data, including study exit data
* Able and willing to provide adequate locator information for study retention purposes
* Sexually active (at least one coital act in the last 3 months prior to screening)
* HIV negative
* Negative pregnancy test *
* Agree to use a non-barrier form of contraceptive
* Agree to adhere to study visits and procedures

  * breastfeeding is not exclusionary but participants must be informed of the presence of TFV in breast milk in negligible amounts

Exclusion Criteria:

* Has creatinine clearance ,<50ml/min, as estimated using the method of Cockcroft and Gault
* Has any other condition, that based on the opinion of the investigator or designee would preclude provision of informed consent, make participation in the study unsafe, complicate interpretation of the study outcome data, or otherwise interfere with achieving the study objectives

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Overall acceptability | over 3 months of use
  Overall acceptability of user-filled, paper applicator compared to prefilled, plastic applicator
context of use | over three months
  Description of context of use of user-filled, paper applicator
challenges encountered | over three months
  Challenges encountered during use of user-filled, paper applicator and recommendations to address challenges
Applicator Preference | Over three months
  Applicator preferences between the user-filled, paper applicator and prefilled, plastic applicator

CONTACTS AND LOCATIONS:
Overall Officials: Leila E Mansoor, Ph.D., Principal Investigator — Centre for the AIDS Programme of Research in South Africa
Locations (1):
- CAPRISA Vulindlela Clinical Research Site, Pietermaritzburg, KwaZulu-Natal, South Africa